CLINICAL TRIAL: NCT03176199
Title: An Interventional, Open Label, and Randomized Controlled Study to Compare the Titration Efficacy and Safety of Control-released Oxycodone and Immediate-released Oxycodone in Opioid-naive Patients With Moderate to Severe Cancer Pain
Brief Title: A Study to Compare the Titration Efficacy and Safety of Control-released Oxycodone and Immediate-released Oxycodone in Patients With Moderate to Severe Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taiwan Mundipharma Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXY15-TW-401
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Pain
Keywords: control-released oxycodone; immediate-released oxycodone; cancer pain; opioid-naive
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-released oxycodone (Experimental): Control-released oxycodone Q12H, initial daily dose is 20 mg + immediate-released oxycodone for PRN
  Interventions: Drug: Oxycodone
- Immediate-released oxycodone (Active Comparator): Immediate-released oxycodone Q6H, initial daily dose is 20mg + immediate-released oxycodone for PRN
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Every 12 hours for control-released oxycodone (OxyContin®)
  Arms: Control-released oxycodone
Drug: Oxycodone — Every 6 hours for immediate-released oxycodone (OxyNorm®)
  Arms: Immediate-released oxycodone

SUMMARY:
This study is to evaluate the efficacy and safety of a titration method by selects 10 mg control-released (CR) oxycodone tablet as background drug in combined with immediate-released (IR) oxycodone, compared to conventional titration method with immediate-released (IR) oxycodone in patients with moderate to severe cancer pain in Taiwan.

DETAILED DESCRIPTION:
This is an interventional, open label, randomized controlled study carrying in multi-centers. Eighty opioid-naive patients with moderate to severe cancer pain (≥ 4) in outpatient department (OPD), who agreed and signed informed consent will be randomly assigned in a 1:1 ratio to receive CR + IR oxycodone or conventional IR oxycodone groups. The study is to compare the titration efficacy and safety of CR with IR oxycodone (experimental group) comparing IR oxycodone (control group) in cancer patients suffered with moderate to severe pain. The study last 14 days. Patients begin the study by the first day visit of the clinic and received the study medication (Baseline). Following visits on cycle 1 (day 3 or 4 depends on the available clinics), cycle 2 (day 7±1), cycle 3 (day 10±1), and cycle 4 (day 14±1). In the experimental group, 10 mg CR oxycodone tablet will be selected as background dose of titration, and patients will be administered once every 12 hrs. Meanwhile, the titration with IR oxycodone will be added according to the pain intensity, e.g. if patient receiving 6 tablets of 10 mg CR oxycodone (giving in Q12H frequency for 3 days), 12 capsules of 5mg IR oxycodone will be dispensed for managing acute pain (rescue use) for the first cycle. In the control group, the conventional titration with IR oxycodone will be conducted according to pain intensity, using 5 mg as initial dose, e.g. 12 capsules of 5mg IR oxycodone (giving in Q6H frequency for 3 days), 12 capsules of 5mg IR oxycodone will be dispensed for rescue use upon to the first cycle. Patient will record their pain score (4 times in Q6H frequency and before taking the drug), 24hr total dose (total tablets/capsule number), number of breakthrough pain and PRN time and dosage used onto the patient diary. The background dose of each patient will be titrated after cycle 1 by investigators. Titration cycles will be recorded and evaluated pain assessments on cycle 2 (day 7±1), cycle 3 (Day 10±1), cycle 4 (day 14±1). During study, the study nurse will follow patient's daily records, drug use condition every second day by telephone or other contact methods to keep close monitor of patient's condition. The telephone contact for cycle 1 and cycle 3 is acceptable for this study. If the telephone contact is conducted for patient, the 1-week quantities of oxycodone should be dispensed to patient.

The safety for individual patient will be followed during study up to end of treatment (EOT) or early termination (ET). All adverse events (AE(s)) and serious adverse events (SAE(s)) occurred during the study period will be followed until resolution or the event is considered stable.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 20 years old and over
2. Patients with background cancer pain more than or equal to NRS 4 during previous 24 hours, or receive more than or equal to 3 times/day for breakthrough pain medication management
3. ECOG ≤ 2
4. Opioid-naive patients who are not administrated any strong opioid for at least one month prior to the index treatments, who currently with poor pain control and intended to be treated for pain relief with strong opioids. The FDA identifies opioid-naive as who not receiving the following treatment for a week or longer of strong opioids:

1) ≥ 60 mg of morphine daily 2) ≥25 mcg transdermalfentanyl/hour 3) ≥ 8 mg of oral hydromorphone daily or 4) an equianalgesic dose of another opioid

5) Patients who will not be treated with radiotherapy within 7 days prior to randomization and during study

6) Patients who need chemotherapy, long term administration of hormone, targeted therapy, or bisphosphonates therapy should undergo a stable anti-tumor therapy prior to randomization.

7) Patients or his/her caregivers who are able to fill out the diary and questionnaire forms

Exclusion Criteria:

1. Patients diagnosed with non-cancer pain or unexplained pain
2. Patients suffered with post-op pain
3. Patients who cannot be applicable for oral administration
4. Patients who have severe constipation defined by CTCAE grade 3 and above
5. Patients with any disease that may easily lead to respiratory depression
6. Monoamine oxidase inhibitor (MAOI) was administrated one week before randomization
7. There are abnormal lab results, with obvious clinical significance, such as the creatinine ≥ 2 fold of upper limit of normal value, or ALT or AST ≥ 2.5 fold of upper limit of normal value (≥ 5 fold, to the patients with liver metastasis or primary liver cancer), or liver function of Child C grade
8. Patients who have potential risk for surgical operation, which may lead to gastrointestinal stenosis, blind loop or gastrointestinal obstruction; or patient is unable to effectively absorb oral medication through gastrointestinal tract
9. Patients who are drug or alcohol abuse
10. Patients with moderate to severe psychiatric problems
11. Patients who have hypersensitivity to oxycodone
12. Patients who are pregnant or lactating
13. Patients who are clinically unstable or have a life expectancy of less than three months making completion of the trial unlikely

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the variable change of NRS pain score and the number of breakthrough pain to obtain pain control after treatment | Up to 14 days
  The change from baseline of NRS pain score and the daily number of breakthrough pain

SECONDARY OUTCOMES:
To evaluate the percentage of patients in each titration cycle | Up to 14 days
  The percentage of patients in each titration cycle
To evaluate the number of patients who switched/discontinued therapy due to serious adverse events or lack of pain control | Up to 14 days
  The number of patients who switched/discontinued therapy due to serious adverse events or lack of pain control
The total opioid taken within 24hrs daily from baseline to day 14 | Up to 14 days
  The total opioid taken within 24 hrs daily from baseline to day 14
To evaluate the mean daily NRS score of subjects from baseline to day 14 | Up to 14 days
  Mean daily NRS score of patients from baseline to day 14
To evaluate the total daily rescue dose taken (immediate-released oxycodone capsule) for treatment of breakthrough pain among patients from baseline to day 14 | Up to 14 days
  The total daily rescue dose taken (immediate-released oxycodone capsule) for treatment of breakthrough pain among patients from baseline to day 14
To evaluate the tolerability and safety of Oxycodone CR and IR in cancer pain patient | Up to 28 days
  The occurrence rate of adverse events and physical examination status
To evaluate the change from baseline in questionnaire | Up to 14 days
  The change from baseline in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Hung, MSc, Principal Investigator — Taichung Veterans General Hospital
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Chang-hua
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mercadante S, Porzio G, Ferrera P, Fulfaro F, Aielli F, Ficorella C, Verna L, Tirelli W, Villari P, Arcuri E. Low morphine doses in opioid-naive cancer patients with pain. J Pain Symptom Manage. 2006 Mar;31(3):242-7. doi: 10.1016/j.jpainsymman.2006.01.001. PMID 16563318
- [Background] Mercadante S. Opioid titration in cancer pain: a critical review. Eur J Pain. 2007 Nov;11(8):823-30. doi: 10.1016/j.ejpain.2007.01.003. Epub 2007 Feb 28. PMID 17331764
- [Background] Klepstad P, Kaasa S, Jystad A, Hval B, Borchgrevink PC. Immediate- or sustained-release morphine for dose finding during start of morphine to cancer patients: a randomized, double-blind trial. Pain. 2003 Jan;101(1-2):193-8. doi: 10.1016/s0304-3959(02)00328-7. PMID 12507714
- [Background] Ripamonti CI, Santini D, Maranzano E, Berti M, Roila F; ESMO Guidelines Working Group. Management of cancer pain: ESMO Clinical Practice Guidelines. Ann Oncol. 2012 Oct;23 Suppl 7:vii139-54. doi: 10.1093/annonc/mds233. No abstract available. PMID 22997447
- [Background] Caraceni A, Hanks G, Kaasa S, Bennett MI, Brunelli C, Cherny N, Dale O, De Conno F, Fallon M, Hanna M, Haugen DF, Juhl G, King S, Klepstad P, Laugsand EA, Maltoni M, Mercadante S, Nabal M, Pigni A, Radbruch L, Reid C, Sjogren P, Stone PC, Tassinari D, Zeppetella G; European Palliative Care Research Collaborative (EPCRC); European Association for Palliative Care (EAPC). Use of opioid analgesics in the treatment of cancer pain: evidence-based recommendations from the EAPC. Lancet Oncol. 2012 Feb;13(2):e58-68. doi: 10.1016/S1470-2045(12)70040-2. PMID 22300860
- [Background] Pan H, Zhang Z, Zhang Y, Xu N, Lu L, Dou C, Guo Y, Wu S, Yue J, Wu D, Dai Y. Efficacy and tolerability of oxycodone hydrochloride controlled-release tablets in moderate to severe cancer pain. Clin Drug Investig. 2007;27(4):259-67. doi: 10.2165/00044011-200727040-00005. PMID 17358098
- [Background] Salzman RT, Roberts MS, Wild J, Fabian C, Reder RF, Goldenheim PD. Can a controlled-release oral dose form of oxycodone be used as readily as an immediate-release form for the purpose of titrating to stable pain control? J Pain Symptom Manage. 1999 Oct;18(4):271-9. doi: 10.1016/s0885-3924(99)00079-2. PMID 10534967